CLINICAL TRIAL: NCT06287619
Title: Post-operative Intravenous Iron to Treat Iron-deficiency Anemia in Patients Undergoing Cardiac Surgery: A Pilot, Multi-centre, Placebo-controlled Randomized Trial.
Brief Title: Post-operative Intravenous Iron to Treat Iron-deficiency Anemia in Patients Undergoing Cardiac Surgery
Acronym: POAM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Kingston Health Sciences Centre (Other); Sunnybrook Health Sciences Centre (Other); Heart and Stroke Foundation of Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22-5685
Record Dates: First submitted 2024-02-23; First posted 2024-03-01 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-06

CONDITIONS: Chronic Iron Deficiency Anaemia; Cardiac Surgery
Keywords: Ferric derisomaltose (Monoferric); Intravenous Iron
MeSH Terms: interventions — ferric derisomaltose; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: POAM is a multicenter, randomized, controlled, internal pilot trial, using a conventional, parallel group, two-armed design at 3 cardiac surgery centres in Canada.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a blinded study, with patients randomized to receive ferric derisomaltose (Monoferric) or placebo. Given that the products have different physical appearances, an unblinded research pharmacist/delegated staff will prepare the IMP then blind the appearance of the IMP for both the intervention group and control group by covering the IV bag and tubing with opaque plastic. All other clinicians, research coordinators, outcome assessors, and patients will remain blinded by using a generic product label in the patient chart and/or the electronic product name (i.e., POAM study drug dose 1 and dose 2, rather than specifying type of product used).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Patients randomized to the IV iron group will receive 1000 mg ferric derisomaltose (Monoferric) diluted in 100 mL of 0.9 % sodium chloride solution, via intravenous infusion over 1 hour using an opaque IV bag and tubing for blinding.
  Interventions: Drug: Monoferric Injectable Product
- Control group (Placebo Comparator): Patients randomized to the placebo group will receive 100 mL of 0.9 % sodium chloride solution via intravenous infusion using an opaque IV bag and tubing for blinding.
  Interventions: Other: 0.9% sodium chloride solution

INTERVENTIONS:
Drug: Monoferric Injectable Product — Ferric derisomaltose will be prepared by an unblinded research pharmacist/delegated staff as per standard of care procedures. Specifically, 10 mL (containing 1000 mg ferric derisomaltose) will be diluted in 100 mL of sterile 0.9% sodium chloride solution and drawn up into blinded syringes and tubing. The 1000 mg doses of ferric derisomaltose will be administered by a bedside nurse over 60 minutes via an infusion pump through a dedicated IV.
  Other Names: Ferric derisomaltose
  Arms: Intervention Group
Other: 0.9% sodium chloride solution — Patients in the control group will receive placebo, which will be 100 mL of sterile 0.9% sodium chloride solution and drawn up into blinded syringes and tubing according to good manufacturing practice (GMP).
  Arms: Control group

SUMMARY:
POAM is a multicenter, randomized, controlled, internal pilot trial, using a conventional, parallel group, two-armed design at 3 cardiac surgery centres in Canada. The study is designed to assess the feasibility of a future, definitive RCT investigating whether, in patients with chronic iron-deficiency anemia undergoing cardiac surgery, IV iron therapy in the postoperative period (initiated shortly after surgery, and repeated at 42 days after surgery, if needed) improves clinical outcomes (days alive and out of hospital at 90 days after surgery; DAOH-90) relative to placebo.

ELIGIBILITY:
Inclusion Criteria:

Patients who are undergoing any non-emergency open cardiac surgery and who meet all following criteria:

1. Age greater than 18 years old
2. Preoperative iron-deficiency with or without anemia (defined as Hb <130 g/L) with any one of:

   1. ferritin ≤100 μg/l; or
   2. ferritin ≤ 300 μg/L and transferrin saturation ≤ 20%; or
   3. reticulocyte Hb content < 29 pg, where available

Exclusion Criteria:

Patients who meet any of the following criteria are not eligible for the study:

1. specialized procedures (e.g., ventricular assist device insertion, thoracoabdominal aneurysm, complex adult congenital surgery and heart transplant)
2. established contraindications to IV iron:

   1. hypersensitivity to the iron product
   2. history of >2 food and/or drug allergic reactions (excluding drug intolerance)
   3. non-iron deficiency anemias such as myelodysplastic syndrome
   4. history of iron overload or disturbances in use of iron such as hemochromatosis or hemosiderosis
   5. decompensated liver cirrhosis (MELD ≥ 19) or active hepatitis
   6. active infection
3. preoperative unstable hemodynamics defined as the requirement for vasopressors or inotropes, or active bleeding (as noted in the clinical record and/or defined as a requirement for red blood cell transfusion for ongoing clinical bleeding)
4. refusal of blood products for religious or other reasons
5. known pregnancy
6. already enrolled in this trial
7. enrolment in another interventional trial which may impact anemia or transfusion management (for example, a trial of hemostatic therapies, such as tranexamic acid)
8. receipt of intravenous iron at any point in the 6 weeks prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility Outcome 1: Percentage of major protocol deviations | through study completion, an average of 1 year.
  Percentage of major protocol deviations with a feasibility threshold of ≤ 5% (i.e., treatment not according to randomization allocation or dosing schedule; treatment initiated in ineligible patients or outside of allotted periods)
Feasibility Outcome 2: Adequate patient enrollment | through study completion, an average of 1 year.
  Adequate patient enrollment defined as ≥20% of eligible patients enrolled.
Feasibility Outcome 3: Percentage of patients lost to follow-up at 90 days | through study completion, an average of 1 year.
  Percentage of patients lost to follow-up at 90 days with a feasibility threshold of ≤ 5%.

CONTACTS AND LOCATIONS:
Overall Officials: Justyna Bartoszko, MD, Principal Investigator — University Health Network, Toronto; Jeannie Callum, MD, Principal Investigator — Kingston Health Sciences Centre; Yulia Lin, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (3):
- Canada (3):
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Toronto General Hospital - University Health Network, Toronto, Ontario

REFERENCES:
- [Derived] Bartoszko J, Miles S, Ansari S, Grewal D, Li M, Callum J, McCluskey SA, Lin Y, Karkouti K. Postoperative intravenous iron to treat iron-deficiency anaemia in patients undergoing cardiac surgery: a protocol for a pilot, multicentre, placebo-controlled randomized trial (the POAM trial). BJA Open. 2024 Jul 27;11:100303. doi: 10.1016/j.bjao.2024.100303. eCollection 2024 Sep. PMID 39161801